CLINICAL TRIAL: NCT01278589
Title: Acute Effect of Plantago Asiatica L. Extract on Antioxidative Biomarkers in Subjects With Mild Hyperlipidemia: A Pilot Study
Brief Title: Antioxidative Effect of Plantago Asiatica L. Extract
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ewha Womans University (Other)
Collaborators: Ministry for Food, Agriculture, Forestry and Fisheries, Korea (Other Government)
Responsible Party: Principal Investigator, Oran Kwon, Ph.D, Professor, Ewha Womans University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: PLA_Biofood
Record Dates: First submitted 2011-01-18; First posted 2011-01-19 (Estimated); Last update posted 2011-10-28 (Estimated); Status verified 2011-10

CONDITIONS: Oxidative Stress

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- • Plantago asiatica L. extract 5g (Experimental)
  Interventions: Dietary Supplement: Plantago asiatica L. extract 5g
- Plantago asiatica L. extract 10g (Experimental)
  Interventions: Dietary Supplement: Plantago asiatica L. extract 10g
- Plantago asiatica L. extract 20g (Experimental)
  Interventions: Dietary Supplement: Plantago asiatica L. extract 20g
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Plantago asiatica L. extract 5g — Liquid (80g) containing Plantago asiatica L. extract 5g
  Arms: • Plantago asiatica L. extract 5g
Dietary Supplement: Plantago asiatica L. extract 10g — Liquid (80g) containing Plantago asiatica L. extract 10g
  Arms: Plantago asiatica L. extract 10g
Dietary Supplement: Plantago asiatica L. extract 20g — Liquid (80g) containing Plantago asiatica L. extract 20g
  Arms: Plantago asiatica L. extract 20g
Dietary Supplement: Placebo — Liquid (80g) without Plantago asiatica L. extract
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the antioxidant effect of Plantago asiatica L. extract in subjects with mild hyperlipidemia.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate an acute effect of Plantago asiatica L. extract consumption on antioxidative biomarkers in subjects with mild hyperlipidemia. Subjects will intake Plantago asiatica L. extract with a high fat meal for oxidative stress loading. Antioxidative biomarkers will be measured after single-dose administration of Plantago asiatica L. extract.

ELIGIBILITY:
Inclusion Criteria:

* Adults age over 30
* BMI(Body mass index) between 25 and 33 kg/m2
* Total cholesterol between 200mg/dL and 250mg/dL OR Triglyceride between 150mg/dL and 220mg/dL OR LDL-cholesterol between 130mg/dL and 165mg/dL

Exclusion Criteria:

* Subject who has taken part in other clinical trials within 30 days of screening visit
* Subject who has taken medicines, Chinese medicines and Health/Functional Foods which can affect antioxidative biomarkers within 30days of screening visit
* Subject who is pregnant or breast feeding
* Subject who lost body weight over 4kg within 30days of screening visit
* Alcoholic
* Smoker
* Subject who takes excessive exercise (over 7hours/week)
* Subject who has hypertension(≥140/90mmHg), diabetes(fasting blood glucose ≥126mg/dL), kidney disease, hepatic disease or hyperthyroidism within 2years
* Subject who has an allergy to the ingredients of study product

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-12; Primary Completion 2011-04 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Comet assay after single-dose consumption of Plantago asiatica L. extract | measured 5 times over 6 hours(0, 60, 120, 240, 360 minutes)

SECONDARY OUTCOMES:
Plasma FRAP | measured 5 times over 6 hours(0, 60, 120, 240, 360 minutes)
Plasma MDA | measured 5 times over 6 hours(0, 60, 120, 240, 360 minutes)
Plasma FFA | measured 5 times over 6 hours(0, 60, 120, 240, 360 minutes)
Plasma ox-LDL | measured 5 times over 6 hours(0, 60, 120, 240, 360 minutes)
Plasma erythrocyte SOD | measured 5 times over 6 hours(0, 60, 120, 240, 360 minutes)
Plasma triglyceride | measured 5 times over 6 hours(0, 60, 120, 240, 360 minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Oran Kwon, Ph.D, Principal Investigator — Ewha Womans University
Locations (1):
- Ewha Womans University / Hanaro Medical Foundation, Seoul, South Korea

REFERENCES:
- [Background] Sun Y. Free radicals, antioxidant enzymes, and carcinogenesis. Free Radic Biol Med. 1990;8(6):583-99. doi: 10.1016/0891-5849(90)90156-d. PMID 2193855
- [Background] Liu X, Wu X, Huang H, Zhong S, Lai X, Cao L. [Herbalogical study on Plantago asiatica L]. Zhong Yao Cai. 2002 Jan;25(1):46-8. Chinese. PMID 12583244
- [Background] Choi SY, Jung SH, Lee HS, Park KW, Yun BS, Lee KW. Glycation inhibitory activity and the identification of an active compound in Plantago asiatica extract. Phytother Res. 2008 Mar;22(3):323-9. doi: 10.1002/ptr.2316. PMID 18167045
- [Background] Chung MJ, Park KW, Kim KH, Kim CT, Baek JP, Bang KH, Choi YM, Lee SJ. Asian plantain (Plantago asiatica) essential oils suppress 3-hydroxy-3-methyl-glutaryl-co-enzyme A reductase expression in vitro and in vivo and show hypocholesterolaemic properties in mice. Br J Nutr. 2008 Jan;99(1):67-75. doi: 10.1017/S0007114507798926. Epub 2007 Aug 15. PMID 17697428
- [Background] Xu C, Luo L, Tan RX. Antidepressant effect of three traditional Chinese medicines in the learned helplessness model. J Ethnopharmacol. 2004 Apr;91(2-3):345-9. doi: 10.1016/j.jep.2004.01.012. PMID 15120459
- [Background] Lee SJ. Korean folk medicine. Publishing center of Seoul National Unicersity, Seoul. P 130, 1966
- [Background] Jeong CH, Bae YI, Shim KH, Choi JS. DPPH radical scavenging effect and antimicrobial activities of Plantain (Plantago asiatica L.) extracts. J Korean Soc Food Sci Nutr 33(10): 1601-1605, 2004